CLINICAL TRIAL: NCT01199835
Title: The Effects of Dairy Products on Energy Balance
Acronym: MEPEB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Collaborators: The Ministry of Science, Technology and Innovation, Denmark (Other Government); The Danish Dairy Research Foundation, Denmark (Other)
Responsible Party: Principal Investigator, Arne Astrup, Department of Human Nutrition, University of Copenhagen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: B251
Record Dates: First submitted 2010-09-08; First posted 2010-09-13 (Estimated); Last update posted 2014-06-11 (Estimated); Status verified 2014-06

CONDITIONS: Obesity
Keywords: obesity; metabolic syndrome; fecal fat excretion; fecal calcium; weight loss; appetite regulation; intestinal micro flora; lipid profile; energy balance
MeSH Terms: conditions — Obesity; Metabolic Syndrome; Weight Loss

ARMS (2):
- high calcium (Experimental): Dietary intake of calcium ~ 1500 mg/ d, including ~1200 mg/d from dairy products
  Interventions: Other: High Calcium intake from dairy products
- Low calcium (Active Comparator): Low dietary intake of calcium, i.e. ~ <600 mg/d, including 0-1 portion of dairy products
  Interventions: Other: High Calcium intake from dairy products

INTERVENTIONS:
Other: High Calcium intake from dairy products — High dietary intake of calcium from dairy products (~1200 mg/d)

SUMMARY:
The aim of the study is to investigate the long time effects of high and low intake of dairy products on fecal fat excretion, weight loss, blood pressure, lipid profile, lipid oxidation and appetite regulation in moderately overweight men and women over 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

* men and women,
* medium overweight (body mass index 28-36 kg/m2),
* 18-60 years old,
* low habitual calcium intake (<800 mg/d)

Exclusion Criteria:

* milk allergy, infection diseases and diabetes,
* intake of dietary supplements,
* smoking,
* pregnancy and/or breast feeding,
* any medications known to affect the outcome measurements,
* weigh reducing diet,
* gastrointestinal diseases,
* participation in other intervention studies

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2010-06; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Fecal fat excretion | 24 weeks
Body weight | 24 weeks
body composition | 24 weeks

SECONDARY OUTCOMES:
Resting energy expenditure | 24 weeks
Blood pressure | 24 weeks
Appetite regulation | 24 weeks
Lipid profile | 24 weeks
Intestinal micro flora | 24 weeks
Metabolomics in urine, feces and blood | 24 week
calcium excretion | 24 weeks
bone markers | 24 weeks
vitamin D status | 24 weeks
calcium status | 24 weeks
lipid metabolism | 24 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Exercise, Nutrition and Sports, Faculty of Sciences, University of Copenhagen, Frederiksberg, Denmark